CLINICAL TRIAL: NCT00699478
Title: Effect of Oral Vitamin B12 Administration for Vitamin B12 Deficiency After Total Gastrectomy
Brief Title: Oral Vitamin B12 Administration for Vitamin B12 Deficiency After Total Gastrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Woo Jin Hyung, Associate professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0460
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Vitamin B12 Deficiency
Keywords: vitamin B12 deficiency; post total gastrectomy; stomach cancer
MeSH Terms: conditions — Vitamin B 12 Deficiency; Stomach Neoplasms | interventions — mecobalamin; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): post total gastrectomized patients due to gastric cancer who has vitamin B12 deficiency - given oral vitamin B 12 supplementation
  Interventions: Drug: mecobalamin

INTERVENTIONS:
Drug: mecobalamin — Methycobal Tab 0.5mg (contains 0.5 mg mecobalamin) for 3 times a day (Q8hrs) for three months
  Other Names: actinamide; cobalamin

SUMMARY:
Pernicious anemia develops in 50% of total gastrectomized due to gastric cancer patients. Lack of intrinsic factor, which is secreted by parietal cell from stomach wall causes deficiency of cobalamin, which, in final, causes pernicious anemia. Thus, patients who had undergone total gastrectomy needs to be provided externally with cobalamin. Until now, intramuscular injection of cyanocobalamin has been the choice of treatment for cobalamin deficiency, but it has demerits in that it causes discomfort of coming to the hospital to get an injection, and in its high costs.

However, in pernicious anemia in old age and absorption disorder patients, it has been reported that oral administration of cobalamin had effect of elevating serum vitamin B12. Thus, this study was designed to prove the effect of oral administration of vitamin B12 in total gastrectomized patients with cobalamin deficiency.

DETAILED DESCRIPTION:
Vitamin B 12 is important for hexane synthesis. Its deficiency causes pernicious anemia and abnormal functioning neurons. It is not synthesized intrinsically, and extrinsic supplement is vital. Vitamin B 12 is known to be abundant in meat and dairies. It is usually absorbed in form of cobalamin and forms a complex with R binder, decomposed in duodenum, again form a complex with intrinsic factor, and finally absorbed in terminal ileum.

In this process, intrinsic factor takes a major role, but when total gastrectomized, absorption of cobalamin is impossible theoretically, because intrinsic factor is known to be produced only from mucosa of the stomach. Thus,deficiency of vitamin B 12 develops, which causes clinical symptoms of pernicious anemia and neurological disorders.

Total gastrectomy for cure of upper body cancer of stomach is gradually growing in Korea and Japan, and more than 50% of the patients are reported to have deficiency of vitamin B12. Pernicious anemia and irreversible neurologic disorder can develop, thus supplementing the vitamin is an important treatment for the patient. However, the protocol in supplementation has not been exhibited as yet.

Reported as now in Korea, after average six months postoperation, decrease of vitamin B12 was seen, and it is recommended that injection of Actinamide monthly after six months for supplementation should be the protocol for total gastrectomized patient.

Intramuscular injection of Actinamide is the choice of treatment for vitamin B12 deficiency for total gastrectomized patient. However, having to visit hospital and the high cost of intramuscular vitamin B12 is a big burden for the patients. Van Walraven et al. from Canada reported in 2001, that when comparing the cost for oral supplementation of vitamin B12 with intramuscular injection, the difference of cost could rise up to 2 billion dollars. Oral supplementation of vitamin B12 is simple to use, can lower the number of hospital visits, and lessen the injection related complications, and thus improve the quality of life of the patient and bring reduction of medical expense.

However, effect of oral supplementation of vitamin B12 has not been studied in Korea. In Japan, Adachi et al. has reported that oral supplementation has effects on total gastrectomized patients, although its mechanism was not known.

Studies on oral supplementation of vitamin B12 for total gastrectomized patient are rare, thus this study was aimed to prove the effect of oral vitamin B12 in total gastrectomized patients, and to establish a protocol for postoperation follow up.

ELIGIBILITY:
Inclusion Criteria:

* Undergone total gastrectomy for gastric cancer
* Regular follow up is possible
* Serum vit,. B12 < 200pg/ml

Exclusion Criteria:

* Has diseases other than stomach cancer
* Patients with other kinds of oral supplementation (multi-vitamins)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Serum vitamin B12 | 1,2 and 3 months after administration of medicine

SECONDARY OUTCOMES:
Questionnaire | 1,2,3 months after administration of medicine
MCV | 1,2,3 months after administration of medicine
Serum Homocysteine | 1,2,3 months after administration of medicine
TIBC | 1,2,3 months after administration of medicine
Serum iron | 1,2,3 months after administration of medicine
Transferrin | 1,2,3 months after administration of medicine

CONTACTS AND LOCATIONS:
Overall Officials: Woo Jin Hyung, Ph.D, Principal Investigator — Yonsei University
Locations (1):
- Yonsei university college of medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Bernard M, Babior H., Franklin Bunn. Megaloblastic anemias. In: Dennis LK, Anthony SF, Eugine B, Stephen LH, Dan LL, J.Larry J. editors. Harrison's Principles of internal medicine. 16th ed. New York: Mcgraw-Hill companies; 2005. p.601-7.
- [Background] Tai Il Seo, Sung Joon Kwon:A Study for Incidence and Treatment of Vitamin B12 Deficiency after Total Gastrectomy. J Korean Surg Soc 2003;64:206-11.(In Korean)
- [Background] van Walraven C, Austin P, Naylor CD. Vitamin B12 injections versus oral supplements. How much money could be saved by switching from injections to pills? Can Fam Physician. 2001 Jan;47:79-86. PMID 11212437
- [Background] Oh R, Brown DL. Vitamin B12 deficiency. Am Fam Physician. 2003 Mar 1;67(5):979-86. PMID 12643357
- [Background] Adachi S, Kawamoto T, Otsuka M, Todoroki T, Fukao K. Enteral vitamin B12 supplements reverse postgastrectomy B12 deficiency. Ann Surg. 2000 Aug;232(2):199-201. doi: 10.1097/00000658-200008000-00008. PMID 10903597
- [Background] Hyun Dong Chae, Ki Ho Park. Vitamin B12 Deficiency after a Total Gastrectomy in Patients with Gastric Cancer. Korean Gastric Cancer Assoc 2006;6(1):6-10.(In Korean)